CLINICAL TRIAL: NCT03107416
Title: Phase I/II Study of Transarterial Hepatic Embolization With Bumetanide in Unresectable Hepatocellular Carcinoma
Brief Title: Delivering a Diuretic Into the Liver Artery Followed by Plugging up the Artery to Starve Out Liver Cancer Cells
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-141
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Unresectable Hepatocellular Carcinoma
Keywords: Bumetanide; Diuretic; Transarterial Embolization (TAE); 17-141
MeSH Terms: interventions — Bumetanide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bumetanide (Experimental): Three escalating doses of bumetanide will be used: 0.01 mg/kg (level 1), 0.02 mg/kg (level 2) and 0.04 mg/kg (level 3) in a standard 3+3 design. Starting with level 1, three patients will first be enrolled at each level.
  Interventions: Procedure: Hepatic artery embolization (HAE); Drug: Bumetanide

INTERVENTIONS:
Procedure: Hepatic artery embolization (HAE) — The intervention being studied is HAE for the treatment of HCC in combination with Bumetanide. HAE is a standard of care procedure.
Drug: Bumetanide — Intra-arterial (IA) injection of 0.01mg/kg of Bumetanide in the first cohort, 0.02 mg/kg in the second cohort and 0.04 mg/kg of IA Bumetanide in the final cohort patients during standard HAE until stasis is evident.

SUMMARY:
The purpose of this study is to test the safety of Bumetanide , at different doses to find out what effects, if any, it has on people who undergo tumor TAE as part of their regular care. Bumetanide is a commonly used medication to reduce the amount of water in the body.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnoses of HCC according to European Association for the Study of Liver disease (EASL) criteria for diagnosis (See Appendix 1). Regional lymphadenopathy will be allowed.

  * Any virus status accepted (e.g. Hepatitis C etc.)
  * Any prior liver treatment
* Patients within unresectable HCC
* At least 18 years old
* ECOG performance status 0 or 1
* Radiographically measurable disease per mRECIST 1.1
* Meets standard of care to undergo embolization

Exclusion Criteria:

* Women who are pregnant or lactating
* Documented hypersensitivity to bumetanide or sulfonamides
* Patients with resectable HCC
* High risk for post-embolization hepatic failure:

  °Child's C cirrhosis

  °> 80% liver involvement by tumor
* Contraindication to angiography/embolization including:

  * Patients cannot receive contrast:
  * Severe allergic reaction to contrast despite premedication
  * Poor renal function not on dialysis
  * Other, based on judgment of the investigator
* ECOG score 2
* Main portal vein tumor thrombus
* BCLC D = patients with distant metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2026-04-05 (Estimated); Study Completion 2026-04-05 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) (phase I) | 1 year
  Three escalating doses of bumetanide will be used: 0.01 mg/kg (level 1), 0.02 mg/kg (level 2) and 0.04 mg/kg (level 3) in a standard 3+3 design. Starting with level 1, three patients will first be enrolled at each level.
estimate the local tumor progression (LTP) rates (phase II) | 1 year
  After the last first stage patient has three months followup, 6-month LTP will be estimated using Kaplan-Meier methods. If the one-sided 90% lower confidence bound is less than 40% the study will stop. Otherwise 12 more patients will be enrolled for a total of 30. At the end of the study 12-month LTP will be estimated using competing risk (cumulative incidence) methods.

CONTACTS AND LOCATIONS:
Overall Officials: Hooman Yarmohammadi, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan Kettering Basking Ridge (Consent and follow-up only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent and follow-up only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent and follow-up only), Montvale, New Jersey
  - Memorial Sloan Kettering Westchester (Consent and follow-up only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm